CLINICAL TRIAL: NCT05518461
Title: iThrive WI - A Smartphone Intervention for Overdose and Risk and COVID-19 Among People Who Use Drugs
Brief Title: Smartphone Intervention for Overdose and COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-0956; A545000 (Other: UW Madison); Protocol Version 7/29/2022 (Other: UW Madison); UG3DA044826-01 (NIH); NUR/FACULTY AFFAIRS/ADMIN (Other: UW Madison)
Record Dates: First submitted 2022-08-25; First posted 2022-08-26 (Actual); Results first posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Substance Use Disorders; Overdose; COVID-19
MeSH Terms: conditions — Substance-Related Disorders; Drug Overdose; COVID-19

STUDY DESIGN:
Intervention Model Description: Preliminary outcomes will be measured from 60 participants at baseline (pre-test), followed by a 12-week intervention through the Thrive4Life Connect smartphone application, and re-assessment of outcomes at months 3 and 6.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iThrive WI Intervention (Experimental): Participants will receive COVID-19 and overdose-related educational and motivational content over the course of 12 weeks through the Thrive4Life Connect, a mobile health application. They will be invited to set goals for lowering overdose and COVID-19 risk.
  Interventions: Device: iThrive WI Intervention

INTERVENTIONS:
Device: iThrive WI Intervention — Participants will receive COVID-19 and overdose-related educational and motivational content over the course of 12 weeks through the Thrive4Life Connect, a mobile health application. They will be invited to set goals for lowering overdose and COVID-19 risk.

SUMMARY:
This study will examine if the use of a smartphone application called Thrive4Life Connect can help people who use drugs lower their risk of overdose and learn more about COVID-19 vaccines. 60 participants will be enrolled and can expect to be on study for up to 6 months.

DETAILED DESCRIPTION:
The mobile health system used in this study, called Thrive4Life Connect, has been developed for use in harm reduction settings with prior funding from the National Institute on Drug Abuse. Thrive4Life Connect is based on the Addiction Comprehensive Health Enhancement Support System (A-CHESS) and facilitates brief, behavioral interventions targeting knowledge gaps, motivation, and social connectedness. This app is being used in another study at University of Wisconsin-Madison (registered to NCT04268173).

The proposed study will develop new intervention content for assessing and increasing vaccine confidence and lowering overdose risk. The feasibility and preliminary efficacy will be tested using a pilot, pre-post study design with 60 people who have injected drugs in the past week and used opioids in the past 30 days. The investigators will examine feasibility outcomes based on study recruitment, retention, and intervention completion. Changes in knowledge about COVID-19 and overdose, motivation to reduce risk, and behavioral outcomes including overdose risk behaviors and vaccine uptake will be examined to establish preliminary efficacy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Willing to attend in person study encounters at any of the following Vivent Health locations: Milwaukee, Appleton, and Eau Claire
* Used opioids to get high in the past 30 days
* Injected drugs at least 2 times in the past 7 days
* Express interest in reducing their overdose risk

Exclusion Criteria:

* None in addition to the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel E Gicquelais, PhD, MPH, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
The plan is to share results in an aggregate format and to not share any data that could be used to identify participants. The investigators will only report summary data to individuals outside the study team and expect to publish manuscripts based on information gathered in this study, but no participants will be identified in these shared results.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | iThrive WI Intervention
Started | 60
Completed at 3 Months | 44
Completed at 6 Months | 38
Completed All 3 Surveys | 35
Completed Only Baseline and 3 Month | 9
Completed Only Baseline and 6 Month | 3
Completed | 35
Not Completed | 25
Not completed — Lost to Follow-up | 25

BASELINE CHARACTERISTICS:
Arm/Group | iThrive WI Intervention
Number analyzed (Participants) | 60
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 34 [29 to 41]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 51
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 47
  More than one race | 4
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Content Completion Rate Assessed as Number of Participants Who Completed at Least 6 of the 12 Weeks of the Intervention
Description: Study feasibility will be in part based on intervention content completion rates. The study will be considered feasible if participants complete any intervention content on at least 50% (i.e., 6) of the 12 weeks. We will report the number of participants who completed at least 6 of the 12 weeks.
Time Frame: up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | iThrive WI Intervention
Number analyzed (Participants) | 60
Participants | 40

2. Secondary Outcome: Number of Days in the Past Month Endorsing Overdose Risk Behaviors
Description: Preliminary effectiveness will in part be measured by examining the number of days in the previous month endorsing overdose risk behaviors at months 3 and 6 (relative to baseline/study enrollment). Overdose risk behavior frequency will be assessed by participant self-report.
Time Frame: baseline, 3 months, 6 months
Population: Losses to follow-up occurred across study measurement timepoints.
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- Non-Injection Opioid Use: Average of the reported number of days of using opioid painkillers, smoking opioids, and snorting opioids within the past 30 days.
- Using Opioids or Stimulants While Alone: Average of the number of days opioids and stimulants were used while alone in the past 30 days.
- Injection Drug Use and/or Speedballing: Average of the reported number of days of opioid injection, stimulant injection, opioid and stimulant use within a 6-hour time periods, and opioid and stimulant use at the same time within the past 30 days.
- Opioid and Alcohol Use: Number of days that opioids and alcohol were used within a 6-hour time frame in the past 30 days.
- Opioid and Benzodiazepine Use: Number of days that opioids and benzodiazepines were used within a 6-hour time frame in the past 30 days.
Arm/Group | Non-Injection Opioid Use | Using Opioids or Stimulants While Alone | Injection Drug Use and/or Speedballing | Opioid and Alcohol Use | Opioid and Benzodiazepine Use
Number analyzed (Participants) | 59 | 57 | 59 | 60 | 58
days
  baseline: number analyzed (Participants) | 53 | 54 | 57 | 57 | 56
  baseline | 2 [0 to 10] | 5 [0 to 15] | 14 [9 to 23] | 0 [0 to 1] | 0 [0 to 0]
  3 months: number analyzed (Participants) | 41 | 41 | 44 | 41 | 41
  3 months | 0 [0 to 3] | 3 [0 to 10] | 9 [4 to 16] | 0 [0 to 0] | 0 [0 to 0]
  6 months: number analyzed (Participants) | 33 | 33 | 34 | 35 | 34
  6 months | 0 [0 to 7] | 1 [0 to 7] | 5 [1 to 16] | 0 [0 to 0] | 0 [0 to 0]

3. Secondary Outcome: Change in COVID-19 Vaccination Rates From Baseline
Description: Preliminary effectiveness will in part be assessed by measuring the proportion of participants vaccinated against COVID-19 at baseline and at months 3 and 6.
Time Frame: baseline, 3 months, 6 months
Population: Losses to follow-up occurred at months 3 and 6, resulting in a different subgroup of participants included in each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | iThrive WI Intervention
Number analyzed (Participants) | 60
Participants
  baseline: number analyzed (Participants) | 59
  baseline | 30
  3 months: number analyzed (Participants) | 38
  3 months | 16
  6 months: number analyzed (Participants) | 33
  6 months | 17

ADVERSE EVENTS:
Time Frame: up to 6 months
Arm/Group | iThrive WI Intervention
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-08): https://cdn.clinicaltrials.gov/large-docs/61/NCT05518461/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-24): https://cdn.clinicaltrials.gov/large-docs/61/NCT05518461/ICF_001.pdf